CLINICAL TRIAL: NCT03919370
Title: Detection of Cerebral Ischemia With Artificial Intelligence- Biomarkers as Indicators in Controlled Cerebral Ischemia and Reperfusion.
Brief Title: Detection of Cerebral Ischemia With Artificial Intelligence.
Acronym: CIDAI-BAS
Status: Completed | Type: Observational
Sponsor: Linda Block (Other)
Collaborators: Göteborg University (Other)
Responsible Party: Sponsor-Investigator, Linda Block, Doctor, MD, PhD, Göteborg University
Organization: Göteborg University (Other)
Other Study IDs: CIDAI-BAS
Record Dates: First submitted 2019-04-05; First posted 2019-04-18 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Ischemia, Cerebral; Ischemic Stroke; Artery Occlusion; Artery Carotid Stenosi; Anesthesia; Surgery
MeSH Terms: conditions — Brain Ischemia; Ischemic Stroke; Arterial Occlusive Diseases; Carotid Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cerebral ischemia: Patients undergoing planned surgery for carotid stenosis
  Interventions: Other: No intervention
- Reperfusion: Patients undergoing cerebral trombectomy.
  Interventions: Other: No intervention
- Anaesthesia and surgery: Patients without preexisting cerebral injury undergoing abdominal surgery and anaesthesia
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — there will be NO intervention

SUMMARY:
In patients undergoing planned surgery for carotid tromendarterendectomy, a non-invasive device that registers heart rate variability is attached. Furthermore a non-invasive device that monitors cerebral oxygenation- near infrared spectroscopy as well as electroencephalography is also attached. At times when surgeons clamps the carotid artery, there will be a moment with controlled cerebral ischemia.

This will be registered by the devices. The information obtained will be used to teach artificial intelligence what patterns are related to cerebral ischemia. The same procedure will be performed in patients undergoing ocklusive cerebral trombectomy, so the artificial intelligence will learn to recognize cerebral reperfusion.Blood samples will be drawn before and after cerebral ischemia may occur and will be analyzed for neurobiomarkers and cardiac biomarkers. To teach the algorithm patterns from anaesthesia and surgery in patients without pre existing neuronal injury, the same method will be applied to patients undergoing mixed abdominal surgery. This group will provide a better knowledge of neuro biomarker patterns during anesthesia and surgery.

DETAILED DESCRIPTION:
The neurobiomarkers that will be analyzed for detection of cerebral ischemia is Glial Fibrillary Acidic Protein, Neurofilament light chains, S-100B, Neuron specific endolas, Total-tau. Cardiac biomarkers are troponin-t and NT-pro brain natriuretic peptide.

Blood sampling will occur before anesthesia induction and 2 and 24 hours after surgery or plausible ischemia for patients undergoing surgery for carotid endarterectomy. For patients undergoing acute thrombectomy blood sampling will be performed as soon as possible after the patient has arrived to the hospital as well as 2 hours and 24 hours later. For patients undergoing mixed abdominal surgery, sampling will be done before anesthesia induction and 2 hours and 24 hours after surgery.

Additionally, blood from the thrombectomy cohort and the control cohort will be analyzed by an external party OLIMK, Uppsala. This is an explorative study aiming to find new biomarkers for detection of cerebral ischemia. Blood from both cohorts will be analyzed for 384 neurology biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Patients planned for carotid surgery or trombectomy
* Giving informed consent to participate

Exclusion Criteria:

* Patients that do not consent Patients with arrythmia or pacemaker

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: See above
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Heart Rate variability | 2020-2030
  Changes in Heart Rate Variability from baseline.
Near infrared spectroscopy | 2020-2030
  Changes in Near Infrared spectroscopy from baseline.
Electroencephalography | 2020-2030
  Changes in electroencephalography from baseline, more precisely the Power in alpha bands, beta band, delta bands and quotas between these.
Biomarkers indicating cerebral ischemia in blood | 2020-2030
  Changes in levels of biomarkers in blood from baseline. Total tau, neurofilament light chains, glial fibrillary acidic protein, S-100, neuron specific endolas.
Biomarkers indicating cardiac ischemia in blood | 2020-2030
  Changes in levels of biomarkers in blood from baseline. Troponin T

CONTACTS AND LOCATIONS:
Overall Officials: Linda Block, PhD, Principal Investigator — Inst Clin Sciences
Locations (1):
- Sahlgrenska University hospital, Gothenburg, Sweden, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Block L, El-Merhi A, Liljencrantz J, Naredi S, Staron M, Odenstedt Herges H. Cerebral ischemia detection using artificial intelligence (CIDAI)-A study protocol. Acta Anaesthesiol Scand. 2020 Oct;64(9):1335-1342. doi: 10.1111/aas.13657. Epub 2020 Jul 2. PMID 32533722